CLINICAL TRIAL: NCT06288139
Title: Management of Open Fracture Tibia in Teenagers in Assiut University Hospital .
Brief Title: Management of Open Fracture Tibia in Teenagers
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mena Rashad Fawzy, Resident doctor, Assiut University
Other Study IDs: open fracture tibia
Record Dates: First submitted 2024-02-21; First posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Open tíbia Fracture

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to study the incidence of open tibial fractures in early teenagers and evaluate the management outcomes

DETAILED DESCRIPTION:
Tibial fractures are the third most common long bone fracture after the femur and forearm, representing 15% of all pediatric fractures Tibial fracture is a common injury in children, and it usually involves the diaphysis and distal metaphyseal region Open fracture tibia must be considered orthopedic emergencies due to the high risk of contamination, osteomyelitis, malformation, nonunion, and disability The anteromedial aspect of the tibia is subcutaneous with no overlying musculature for protection and the middle/distal tibia has no muscular origins, which can delay union in these areas The biology of the repair of fractures in children differs from that in adults in several ways. The soft tissues have excellent healing capacity, uncontaminated devitalised bone is salvageable and periosteum in children can regenerate bone in the presence of bone loss. Union is faster. Modalities of treatment of open fracture tibia in teenagers Including Closed reduction followed by a well- molded casting ,debridement followed by casting , utilization of external fixator (EF) remains a popular choice for open injuries, Severely comminuted and unstable fractures and those with significant soft tissue or vascular injury require external fixation However, pin tract infection (PTI) and refracture are common complications during the application of EF . Elastic Nail has also been reported with an acceptable for the treatment of open tibial fractures

, open reduction and internal fixation (ORIF) was reserved for situations in which an adequate reduction could not be obtained or maintained by conservative, Also Closed reduction and intramedullary nail fixation appropriate for the treatment of extraarticular distal tibial fractures .

ELIGIBILITY:
Inclusion Criteria :

• All patients presenting with isolated open fracture tibia in teenagers (aged 10 to 19 Years old )

Exclusion Criteria:

* Patient who refuse to participate in the study
* Patient less than 10 or more than 19 years old
* Pathologic fractures
* Open Fracture tibia with other bony or organ injury
* Open fracture tibia with soft tissue loss or vascular injury

Ages: 10 Years to 19 Years | Sex: All
Age Groups: Child, Adult
Study Population: All patients fulfilling the inclusion criteria presenting to our hospital during the study period will be included in the study in 2024
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Number | Baseline
  Measure number of teenagers who were admitted to Assiut university hospital with open fracture tibia with the different treatment methodology

SECONDARY OUTCOMES:
To evaluate treatment outcomes | Baseline
  Fracture healing
Soft tissue healing | Baseline
  time taken for soft tissue to be healed
Complication | Baseline
  Incidence and rate of complications

CONTACTS AND LOCATIONS:
Overall Officials: Kamal El gafari, prof, Study Director — Assiut University

REFERENCES:
- [Background] Wang H, Liu H, Wu J, Li C, Zhou Y, Liu J, Ou L, Xiang L. Age, gender, and etiology differences of sports-related fractures in children and adolescents: A retrospective observational study. Medicine (Baltimore). 2019 Jan;98(4):e13961. doi: 10.1097/MD.0000000000013961. PMID 30681556
- [Background] Bartlett CS 3rd, Weiner LS, Yang EC. Treatment of type II and type III open tibia fractures in children. J Orthop Trauma. 1997 Jul;11(5):357-62. doi: 10.1097/00005131-199707000-00010. PMID 9294800
- [Background] Egol KA, Koval KJ, Zuckerman JD. Handbook of Fractures. 5th ed. Philadelphia, USA: Lippincott, Williams and Wilkins; 2015. [Google Scholar]
- [Background] Louie KW. Management of open fractures of the lower limb. BMJ. 2009 Dec 17;339:b5092. doi: 10.1136/bmj.b5092. No abstract available. PMID 20019057
- [Background] Houdek MT, Wagner ER, Wyles CC, Sems SA, Moran SL. Reverse Medial Hemisoleus Flaps for Coverage of Distal Third Leg Wounds: A Technical Trick. J Orthop Trauma. 2016 Apr;30(4):e138-42. doi: 10.1097/BOT.0000000000000491. PMID 26606601
- [Background] Rexiti P, Zhang TC, Batuer C, Cao L. Orthopedic treatment for open fracture of lower extremities and soft tissue defects in young children and rapid rehabilitation after operation. Phys Sportsmed. 2020 May;48(2):161-164. doi: 10.1080/00913847.2019.1642810. Epub 2019 Aug 2. PMID 31317807
- [Background] Charalambous CP, Alvi F, Siddique I, Zenios M, Hirst P, Marshall P. Casting versus surgical fixation for grade IIIA open tibial diaphysial fractures in children: effect on the rate of infection and the need for secondary surgical procedures to promote bone union. Int Orthop. 2005 Dec;29(6):392-5. doi: 10.1007/s00264-005-0009-3. Epub 2005 Aug 10. PMID 16091949
- [Background] Norman D, Peskin B, Ehrenraich A, Rosenberg N, Bar-Joseph G, Bialik V. The use of external fixators in the immobilization of pediatric fractures. Arch Orthop Trauma Surg. 2002 Sep;122(7):379-82. doi: 10.1007/s00402-001-0383-2. Epub 2002 Feb 28. PMID 12228797
- [Background] Dai J, Wang X, Zhang F, Zhu L, Zhen Y. Treatment of distal metaphyseal tibia fractures using an external fixator in children. Medicine (Baltimore). 2019 Sep;98(36):e17068. doi: 10.1097/MD.0000000000017068. PMID 31490405
- [Background] Pandya NK, Edmonds EW. Immediate intramedullary flexible nailing of open pediatric tibial shaft fractures. J Pediatr Orthop. 2012 Dec;32(8):770-6. doi: 10.1097/BPO.0b013e318270468b. PMID 23147618
- [Background] Pandya NK. Flexible Intramedullary Nailing of Unstable and/or Open Tibia Shaft Fractures in the Pediatric Population. J Pediatr Orthop. 2016 Jun;36 Suppl 1:S19-23. doi: 10.1097/BPO.0000000000000754. PMID 27078231
- [Background] Im GI, Tae SK. Distal metaphyseal fractures of tibia: a prospective randomized trial of closed reduction and intramedullary nail versus open reduction and plate and screws fixation. J Trauma. 2005 Nov;59(5):1219-23; discussion 1223. doi: 10.1097/01.ta.0000188936.79798.4e. PMID 16385303